CLINICAL TRIAL: NCT06867978
Title: A Prospective, Multi-Center, Assessor-Blinded Study on the Clinical Efficacy of CCeLL-In Vivo (Confocal Fluorescence Endomicroscopy) for Intraoperative Brain Tumor Diagnosis.
Brief Title: Multi-center Study on CCeLL-In Vivo's Clinical Efficacy for Intraoperative Brain Tumor Diagnosis.
Acronym: PRECISION
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VPIX Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cCeLL_II_2024; Republic of Korea (Other: VPIX Medical Inc.)
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Frozen Sections; Indocyanine Green; Brain Tumor
Keywords: Diagnostic Imaging; intraoperative; confocal laser endomicroscopy
MeSH Terms: conditions — Brain Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This prospective, multicenter, evaluator-blinded clinical trial evaluates the cCeLL - In vivo confocal laser fluorescence microscope for brain tumor diagnosis during surgery.
  Intervention Summary Study Type: Interventional (Diagnostic) Design: Single-group assignment, evaluator-blinded
  Intervention:
  1. ICG injection during surgery
  2. Fluorescence imaging of the tumor margin using cCeLL - In vivo
  3. Comparison with standard frozen and permanent section analyses
  4. Blinded evaluation by pathologists This study aims to enhance tumor margin assessment and improve diagnostic accuracy during brain tumor surgery.
Masking Description: Pathologists will perform diagnoses without access to patient medical records and will not see prior diagnostic results. They will assess tissue samples using only de-identified information, ensuring that fluorescence imaging results do not influence their evaluation. This approach eliminates bias and maintains the integrity of the study's diagnostic comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cCeLL - In vivo Imaging (Experimental): Participants diagnosed with brain tumors will receive an intravenous injection of Indocyanine Green (ICG) during surgery. The cCeLL - In vivo confocal laser fluorescence microscope will be used to capture real-time images of the tumor margins before tissue collection. Standard frozen section and permanent section analyses will then be performed for diagnostic comparison.
  Interventions: Device: cCeLL In vivo; Drug: Indocyanine Green

INTERVENTIONS:
Device: cCeLL In vivo — Dosage Form: Intravenous injection Dosage: 0.1 - 0.5 mg/kg of Indocyanine Green (ICG) Frequency: Single administration during surgery Duration: Real-time imaging performed immediately after ICG injection and used intraoperatively for tumor margin assessment
Drug: Indocyanine Green — fluorescence dye for staining tissue

SUMMARY:
The primary objective of this study is to demonstrate the non-inferiority of cCeLL compared to frozen section analysis. The investigational device is intended for use with indocyanine green (ICG) for fluorescence imaging as an aid in the visualization of vessels (micro- and macro-vasculature) blood flow in the cerebrovascular before, during or after cranial diagnostic and therapeutic procedures, such as tumor biopsy and resection, which is then read and analyzed by trained-professional for intraoperative diagnosis. The comparison will be held by the device with the conventional intraoperative histological frozen section analysis of identical brain tissue samples in the same patient. Both methods will be compared in terms of their accuracy using the standard of practice, the final pathological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* Patients suspected of having a brain tumor who are scheduled for neurosurgery and are considered candidates for tumor resection
* Patients who understand and have signed the informed consent form

The specimens used in this study must meet all of the following criteria:

* Specimens obtained from patients who have agreed to participate in this clinical trial and who meet the inclusion criteria
* Normal tissue specimens obtained unavoidably during tumor resection surgery in tumor patients

Exclusion Criteria:

* Patients undergoing multiple surgeries
* Patients with bacterial or viral infections
* Patients who develop allergic reactions to the investigational medical device
* Patients with a history of allergy to Indocyanine Green (ICG)
* Patients with iodine hypersensitivity
* Patients taking choleretic agents or rifampicin

Specimens meeting any of the following criteria will be excluded from this clinical trial:

- Specimens with unclear tumor presence or carcinoma diagnosis results based on the reference standard permanent section analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-Inferiority of Diagnostic Accuracy (Percentage of Correct Normal/Tumor Classifications) of cCeLL Compared to Frozen Biopsy | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The diagnostic accuracy of cCeLL-In vivo will be assessed by measuring the percentage of correct normal/tumor classifications compared to the reference standard frozen biopsy. Non-inferiority will be determined using pre-specified statistical margins for sensitivity and specificity.

SECONDARY OUTCOMES:
Diagnostic Accuracy, Sensitivity, and Specificity of cCeLL Compared to Frozen Biopsy Across Tumor Types and Locations | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The diagnostic performance of cCeLL-In vivo will be evaluated by calculating accuracy (percentage of correct diagnoses), sensitivity, and specificity across various tumor types and locations. These values will be compared to those obtained using frozen biopsy as the reference standard.
Percentage of Non-Diagnostic Samples in cCeLL Imaging | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The percentage of non-diagnostic samples (images that cannot be used for a definitive diagnosis) obtained using cCeLL-In vivo will be recorded. A lower rate of non-diagnostic samples would indicate higher image usability and reliability.
Time (Minutes) Required to Obtain a Diagnosis Using cCeLL-In vivo vs. Frozen Biopsy Description: | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The time required to obtain a definitive diagnosis will be measured in minutes, from the point of sample collection to the final diagnostic decision. The average diagnostic time for cCeLL-In vivo will be compared to the traditional frozen biopsy method to evaluate potential time efficiency improvements.
Inter-Observer Agreement (Cohen's Kappa Score) Between Two Pathologists Using cCeLL-In vivo Images | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The level of agreement between two independent pathologists interpreting cCeLL-In vivo images will be measured using Cohen's kappa coefficient (κ). The kappa score will quantify inter-observer agreement beyond chance, with values ranging from 0 (no agreement) to 1 (perfect agreement).
Diagnostic Accuracy (Percentage of Correct Tumor Classifications) of AI-Based Brain Tumor Diagnosis Using cCeLL-In vivo Images | Visit 1 (Surgery Day / Intervention Day) as D-Day
  The accuracy of AI-based diagnosis will be measured as the percentage of correct tumor classifications (normal vs. tumor) compared to the reference standard diagnosis made by expert pathologists. Sensitivity, specificity, and overall accuracy will be calculated to evaluate AI performance.

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) may not be shared due to patient privacy concerns, confidentiality agreements, regulatory restrictions, ethical considerations, and institutional policies. Additionally, data protection laws (e.g., GDPR, HIPAA) and proprietary research interests may limit data availability to ensure compliance and safeguard participant information.